CLINICAL TRIAL: NCT02169414
Title: Effect of Three Multiple-dose Regimens of BIA 9 1067 at Steady-state on the Levodopa Pharmacokinetics of a Single-dose of Immediate Release 100/25 mg Levodopa/Carbidopa and 100/25 mg Levodopa/Benserazide in Healthy Subjects
Brief Title: Effect of Three Multiple-dose Regimens of BIA 9 1067 at Steady-state on the Levodopa Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-91067-123
Record Dates: First submitted 2012-01-24; First posted 2014-06-23 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's disease (PD); BIA 9-1067; Opicapone
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; Levodopa; carbidopa, levodopa drug combination; Benserazide; benserazide, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BIA 9-1067 5 mg (Experimental): 1 capsule of 5 mg + 2 capsules of placebo for 18 days levodopa/carbidopa 100/25 mg was administered on Day 11 levodopa/benserazide 100/25 mg was administered on Day 18.
  Interventions: Drug: BIA 9-1067 5 mg; Drug: levodopa/carbidopa 100/25; Drug: Placebo; Drug: levodopa/benserazide 100/25 mg
- BIA 9-1067 15 mg (Experimental): 3 capsules of 5 mg for 18 days levodopa/carbidopa 100/25 mg was administered on Day 11 levodopa/benserazide 100/25 mg was administered on Day 18.
  Interventions: Drug: BIA 9-1067 5 mg; Drug: levodopa/carbidopa 100/25; Drug: levodopa/benserazide 100/25 mg
- BIA 9-1067 50 mg (Experimental): 2 capsules of BIA 9-1067 25 mg + 1 capsule of placebo for 18 days levodopa/carbidopa 100/25 mg was administered on Day 11 levodopa/benserazide 100/25 mg was administered on Day 18.
  Interventions: Drug: BIA 9-1067 25 mg; Drug: levodopa/carbidopa 100/25; Drug: Placebo; Drug: levodopa/benserazide 100/25 mg
- Placebo (Placebo Comparator): 3 capsules of placebo for 18 days levodopa/carbidopa 100/25 mg was administered on Day 11 levodopa/benserazide 100/25 mg was administered on Day 18.
  Interventions: Drug: levodopa/carbidopa 100/25; Drug: Placebo; Drug: levodopa/benserazide 100/25 mg

INTERVENTIONS:
Drug: BIA 9-1067 5 mg — OPC, Opicapone
  Other Names: OPC, Opicapone
  Arms: BIA 9-1067 15 mg; BIA 9-1067 5 mg
Drug: BIA 9-1067 25 mg — OPC, Opicapone
  Other Names: OPC, Opicapone
  Arms: BIA 9-1067 50 mg
Drug: levodopa/carbidopa 100/25 — immediate (standard) release levodopa/carbidopa 100/25
  Other Names: Sinemet®
Drug: Placebo — PLC, Placebo
  Other Names: PLC, Placebo
  Arms: BIA 9-1067 5 mg; BIA 9-1067 50 mg; Placebo
Drug: levodopa/benserazide 100/25 mg — immediate (standard) release levodopa/benserazide
  Other Names: Madopar®

SUMMARY:
The purpose of this study is to determine the effect of BIA 9 1067 (5 mg, 15 mg and 50 mg) in steady-state conditions on the levodopa pharmacokinetics of a single dose of immediate-release levodopa/carbidopa 100/25 mg and of a single dose of immediate-release levodopa/benserazide 100/25 mg.

DETAILED DESCRIPTION:
A single-centre, randomized, double-blind, gender-balanced, placebo-controlled study in 4 groups of 18 healthy subjects each. This study consisted of a once-daily administration of BIA 9 1067 (5 mg, 15 mg or 50 mg) or placebo for 18 days. Twelve (12) hours after the BIA 9 1067 dose, a single-dose of levodopa/carbidopa 100/25 mg was administered on Day 11 and a single-dose of levodopa/benserazide 100/25 mg was administered on Day 18.

ELIGIBILITY:
Inclusion Criteria:

* able to participate and willing to give written informed consent;
* male and female subjects;
* aged 18 to 45 years, inclusive;
* body mass index (BMI) between 18 and 30 kg/m2;
* healthy as determined by the Investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, complete neurological examination and 12-lead electrocardiogram (ECG);
* negative tests for hepatitis B surface (HBs) antigen, anti-hepatitis C virus (HCV), human immunodeficiency virus-1 (HIV-1) and HIV-2 antibodies at screening;
* negative screen for drugs of abuse and alcohol at screening and admission to the treatment period;
* non-smokers or ex-smokers for at least 3 months;
* if sexually active, agreed to use a medically acceptable form of contraception throughout the study;
* if female of childbearing potential, had a negative human chorionic gonadotropin (HCG) beta serum pregnancy test at screening and admission to the treatment period.

Exclusion Criteria:

* who did not conform to the above inclusion criteria, or in case of volunteers who had a clinically relevant surgical history, a clinically relevant family history; or who had a history of relevant atopy;
* who had a significant infection or known inflammatory process at screening or admission to the treatment period; acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, heartburn) at the time of screening or admission to the treatment period;
* who were vegetarians, vegans or had medical dietary restrictions;
* who could not communicate reliably with the Investigator;
* who were unlikely to co-operate with the requirements of the study; history of hypersensitivity to BIA 9 1067, tolcapone, entacapone, levodopa, carbidopa, benserazide or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs;
* any significant cardiovascular (e.g. hypertension), hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidemia), immunologic, dermatological, haematological, neurologic, or psychiatric disease;
* any clinically significant illness in the previous 28 days before day 1 of this study; history of drug abuse within 1 year before study day 1; history of alcoholism within 1 year before day 1.
* Consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g);
* poor motivation, intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements or inability to cooperate adequately, inability to understand and to observe the instructions of the physician;
* donation of blood (i.e., 450 mL) within 60 days before study day 1;
* positive urine screening of ethyl alcohol or drugs of abuse upon admission to the treatment period;
* any history of tuberculosis and/or prophylaxis for tuberculosis; positive results to HIV, hepatitis B surface antigen (HBsAg) or anti-HCV tests;
* participation in any previous clinical study with BIA 9 1067;
* if female, being pregnant or breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BIOTRIAL, Rennes, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg | Placebo
Started | 19 | 19 | 18 | 18
BIA 9-1067 + Levodopa/Carbidopa | 18 | 19 | 18 | 18
BIA 9-1067 + Levodopa/Benserazide | 18 | 18 | 18 | 18
Completed | 18 | 18 | 18 | 18
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg | Total
Number analyzed (Participants) | 18 | 19 | 19 | 18 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 19 | 18 | 74
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 9 | 38
  Male | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration of Levodopa (Levodopa/Carbidopa)
Description: Cmax - Maximum plasma concentration of levodopa following a single oral administration of 100/25 mg levodopa/carbidopa administered 12 h after BIA 9-1067 (5 mg, 15 mg and 50 mg) or placebo on Day 11
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo: 3 capsules of placebo for 18 days levodopa/carbidopa 100/25 mg was administered on Day 11 Levodopa/carbidopa 100/25: immediate (standard) release levodopa/carbidopa 100/25 Placebo: PLC, Placebo
- BIA 9-1067 5 mg: 1 capsule of 5 mg + 2 capsules of placebo for 18 days. Levodopa/carbidopa 100/25 mg was administered on Day 11 BIA 9-1067 5 mg: OPC, Opicapone. Levodopa/carbidopa 100/25: immediate (standard) release levodopa/carbidopa 100/25 Placebo: PLC, Placebo
- BIA 9-1067 15 mg: 3 capsules of 5 mg for 18 days levodopa/carbidopa 100/25 mg was administered on Day 11 BIA 9-1067 5 mg: OPC, Opicapone Levodopa/carbidopa 100/25: immediate (standard) release levodopa/carbidopa 100/25
- BIA 9-1067 50 mg: 2 capsules of BIA 9-1067 25 mg + 1 capsule of placebo for 18 days Levodopa/carbidopa 100/25 mg was administered on Day 11 BIA 9-1067 25 mg: OPC, Opicapone Levodopa/carbidopa 100/25: immediate (standard) release levodopa/carbidopa 100/25 Placebo: PLC, Placebo
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Number analyzed (Participants) | 18 | 18 | 19 | 18
ng/mL | 966.6 (313.2) | 1026.8 (445.2) | 1097.9 (353.2) | 1019.7 (282.1)

2. Primary Outcome: Tmax - Time to Reach Maximum Plasma Concentration of Levodopa (Levodopa/Carbidopa)
Description: Tmax - Time to Reach maximum plasma concentration of levodopa following a single oral administration of 100/25 mg levodopa/carbidopa administered 12 h after BIA 9-1067 (5 mg, 15 mg and 50 mg) or placebo on Day 11
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Number analyzed (Participants) | 18 | 18 | 19 | 18
hours | 0.78 (0.49) | 1 (0.84) | 0.95 (0.55) | 1 (0.59)

3. Primary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve (AUC) of Levodopa From Time Zero to Infinity (Levodopa/Carbidopa)
Description: Levodopa pharmacokinetic parameters following a single oral administration of 100/25 mg levodopa/carbidopa administered 12 h after BIA 9-1067 (5 mg, 15 mg and 50 mg) or placebo on Day 11
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Number analyzed (Participants) | 18 | 18 | 19 | 18
ng.h/mL | 1861.3 (466.5) | 2332.3 (634.9) | 2736.8 (767) | 3182.6 (814.1)

4. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve (AUC) of Levodopa From Time Zero to the Last Sampling Time at Which the Drug Concentration Was at or Above the Lower Limit of Quantification. (Levodopa/Carbidopa)
Description: AUC0-t - Area under the plasma concentration-time curve (AUC) of levodopa from time zero to the last sampling time following a single oral administration of 100/25 mg levodopa/carbidopa administered 12 h after BIA 9-1067 (5 mg, 15 mg and 50 mg) or placebo on Day 11
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Number analyzed (Participants) | 18 | 18 | 19 | 18
ng.h/mL | 1788.3 (461.2) | 2219.7 (616.4) | 2584.3 (794.9) | 2975.9 (799)

5. Primary Outcome: Cmax - Maximum Plasma Concentration of Levodopa (Levodopa/Benserazide )
Description: Levodopa pharmacokinetic parameters following a single oral administration of 100/25 mg levodopa/benserazide administered 12 h after BIA 9-1067 (5 mg, 15 mg and 50 mg) or placebo on Day 18
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo: 3 capsules of placebo for 18 days Levodopa/benserazide 100/25 mg was administered on Day 18. Placebo: PLC, Placebo Levodopa/benserazide 100/25 mg: immediate (standard) release levodopa/benserazide
- BIA 9-1067 5 mg: 1 capsule of 5 mg + 2 capsules of placebo for 18 days Levodopa/benserazide 100/25 mg was administered on Day 18. BIA 9-1067 5 mg: OPC, Opicapone Placebo: PLC, Placebo Levodopa/benserazide 100/25 mg: immediate (standard) release levodopa/benserazide
- BIA 9-1067 15 mg: 3 capsules of 5 mg for 18 days Levodopa/benserazide 100/25 mg was administered on Day 18. BIA 9-1067 5 mg: OPC, Opicapone Levodopa/benserazide 100/25 mg: immediate (standard) release levodopa/benserazide
- BIA 9-1067 50 mg: 2 capsules of BIA 9-1067 25 mg + 1 capsule of placebo for 18 days Levodopa/benserazide 100/25 mg was administered on Day 18. BIA 9-1067 25 mg: OPC, Opicapone Placebo: PLC, Placebo Levodopa/benserazide 100/25 mg: immediate (standard) release levodopa/benserazide
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng/mL | 1770.3 (741.2) | 1379.8 (605.1) | 2118.3 (573.4) | 1813.7 (811.3)

6. Primary Outcome: Tmax - Time to Reach Maximum Plasma Concentration of Levodopa (Levodopa/Benserazide)
Description: as for outcome 5
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Number analyzed (Participants) | 18 | 18 | 18 | 18
hours | 0.89 (0.47) | 1.08 (0.52) | 0.7 (0.3) | 1.08 (0.62)

7. Primary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve (AUC) of Levodopa From Time Zero to Infinity (Levodopa/Benserazide)
Description: as for outcome 5
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng.h/mL | 2360.3 (738.9) | 2660.9 (593.2) | 3655.9 (553.1) | 3979.5 (1406.1)

8. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve (AUC) of Levodopa From Time Zero to the Last Sampling Time at Which the Drug Concentration Was at or Above the Lower Limit of Quantification. (Levodopa/Benserazide)
Description: as for outcome 5
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng.h/mL | 2278.8 (730.4) | 2549.8 (586.6) | 3521.1 (557.7) | 3819.7 (1391.5)

ADVERSE EVENTS:
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 50 mg
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/19 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 3/18 | 12/19 | 9/19 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | BIA 9-1067 5 mg (N=19) | BIA 9-1067 15 mg (N=19) | BIA 9-1067 50 mg (N=18)
Right Peripheral Facial Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | BIA 9-1067 5 mg (N=19) | BIA 9-1067 15 mg (N=19) | BIA 9-1067 50 mg (N=18)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 4 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 5 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other